CLINICAL TRIAL: NCT00675857
Title: A Phase IIa Study of the Safety and Clinical Proof-of-concept of NC-503 (Eprodisate Disodium) in Patients With Type II Diabetes and Features of Metabolic Syndrome
Brief Title: A Phase IIa Proof-of-concept Study of NC-503 in Patients With Type II Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Francis Gauthier, Project Manager, Bellus Health Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-503011
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome X
Keywords: Type II diabetes; Metabolic syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Placebo Comparator)
  Interventions: Other: placebo
- B (Active Comparator)
  Interventions: Drug: NC-503 (eprodisate disodium)

INTERVENTIONS:
Drug: NC-503 (eprodisate disodium) — capsules of 400 mg Dosage: 4 capsules (1600 mg) BID for 26 weeks
  Arms: B
Other: placebo — Dosage: 4 capsules BID for 26 weeks
  Arms: A

SUMMARY:
The main objectives of the current study are to establish the safety and clinical proof-of-concept of NC-503 in inadequately controlled patients with Type 2 diabetes and features of metabolic syndrome treated with either metformin, a sulfonylurea agent, or metformin in combination with a sulfonylurea agent.

DETAILED DESCRIPTION:
Phase IIa Multi-center, randomized, double-blind, placebo-controlled and parallel-designed study.

ELIGIBILITY:
Inclusion Criteria:

* Age and gender eligibility: 30 years and older
* Diagnosis of Type 2 diabetes mellitus
* Patients treated with a stable therapeutic dose of either metformin, a sulfonylurea agent, or metformin in combination with a sulfonylurea agent for a minimum period of 3 months prior to the Screening visit
* Patients must have HbA1C level between 7.0-10.0 %, inclusively at screening
* The participant must have central obesity (Waist circumference) defined per country/ethnic group: Europids: men ≥ 94 cm, women ≥ 80 cm; South Asian, Chinese & Japanese: men ≥ 90 cm, women ≥ 80 cm; and any one of the following metabolic syndrome characteristics at screening:
* Reduced HDL cholesterol ≤ 1.0 mmol/L
* Hypertriglyceridemia ≥ 1.7 mmol/L or treatment for dyslipidemia
* Hypertension: ≥ 130/85 mm Hg blood pressure or treatment with antihypertensive medication.
* Patients must have a Glomerular Filtration Rate (GFR) of ≥ 60 mL/min, and no history of dialysis.

Exclusion Criteria:

* Patients having received insulin, thiazolidinediones (TZDs) or non-thiazolidinedione hypoglycemic agents other than metformin or sulfonylurea agents within three months prior to screening
* Has had, within the last 6 months, evidence of significant heart disease or stroke, including myocardial infarction, unstable angina, coronary bypass and/or percutaneous transluminal coronary angioplasty (PTCA), congestive heart failure (New York Heart Association Class III-IV), or severe ischemic disease
* Patients who have an increased red blood cell (RBC) turn-over or Thalassemia or anemia
* Known HIV or history of viral hepatitis type B or C.
* Any type of diabetes other than Type 2 diabetes
* Significant hepatic enzyme elevation
* Body mass index (BMI) of > 40kg/m2
* Current or previous use of oral or injectable corticosteroids, or conditions that require the use of corticosteroids, during the three months prior to screening

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 26 in HbA1c levels | 26 weeks

SECONDARY OUTCOMES:
Change in HbA1c levels | 26 weeks
The rate of achieving glycemic control | 26 weeks
Change in fasting serum glucose levels | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Chiasson, MD, Principal Investigator — Hotel-Dieu du Centre Hospitalier de l'Université de Montréal
Locations (14):
- Canada (14):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Etobicoke, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Ottawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Laval, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec